CLINICAL TRIAL: NCT06188936
Title: Home Semen Analysis Tests As a Screening Tool for the Initial Assessment of Patients Referred to the Fertility Clinic: Assessing the Feasibility of a Randomised Trial in the UK
Brief Title: Home Semen Analysis Tests As a Screening Tool for Fertility Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Principal Investigator, Ashleigh Holt-Kentwell, Clinical Research Fellow in Reproductive Medicine, University of Aberdeen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2-043-23
Record Dates: First submitted 2023-10-31; First posted 2024-01-03 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: The study consists of three work packages. Work package 1 is a questionnaire to be completed by clinicians and scientists. This concludes their involvement.
  Work package 2 is a survey for patients from which work package 3 participants are recruited - they are able to opt to take part in the subsequent work package at the end of the survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Work Package 1: Survey for clinicians and scientists (Other): Online survey of UK clinicians' and scientists' views on home semen analysis tests, including whether a randomised trial is needed to compare them to standard care, and their willingness to recruit to such a trial.
  Interventions: Other: Survey
- Work package 2: Survey for patients (Other): Sample size: 100 patients. Survey of patients' views prior to undergoing routine laboratory semen analysis, including awareness of home testing.
  Interventions: Other: Survey
- Work package 3: Home testing with ExSeed home semen analysis test and post-test survey (Experimental): Sample size: 25 patients. Assessment of patients' ability to complete home semen testing with the ExSeed® test, opinions on ease of test use, and views after undergoing both laboratory semen analysis and home testing. Results from the ExSeed® test will be compared to the participant's laboratory semen analysis result to assess the accuracy of the home test.
  Interventions: Device: ExSeed®

INTERVENTIONS:
Device: ExSeed® — In work package 3, participants will use the provided ExSeed® device and associated app downloaded onto their smartphone to analyse a semen sample provided at home. The app gives a result of "normal" or "below normal," as well as an exact value for sperm concentration, progressive motility, and total motile sperm count. The patient will send their semen analysis results from the smartphone to the research team via secure email.
  Arms: Work package 3: Home testing with ExSeed home semen analysis test and post-test survey
Other: Survey — Surveys will be completed on a hard copy or electronically.
  Arms: Work Package 1: Survey for clinicians and scientists; Work package 2: Survey for patients

SUMMARY:
Infertility, defined as the inability to conceive after 12 months of regular unprotected intercourse, is estimated to affect 1 in 7 heterosexual couples. Semen analysis, carried out as per the detailed World Health Organisation (WHO) standards in an andrology laboratory, is the primary investigation for the male partner presenting to the fertility clinic and reports on multiple semen parameters. Hospital clinic attendance is required, which could be at a significant distance from the patient's home, to produce a sample at a given appointment time that is then analysed by the laboratory without delay, as the results are time sensitive. A formal report is produced after several weeks. This process was not sustainable during the Covid pandemic and these methods would be threatened by similar situations in the future.

Despite semen analysis being an essential component of fertility work-up the WHO themselves state that the test does not distinguish between fertile and infertile men. In addition, it involves a significant cost to the national healthcare system. Therefore, a more efficient initial test of male fertility warrants consideration.

Home semen analysis tests are a screening tool that provide a simplified, initial assessment. They are widely available to purchase in the UK, but are not currently issued to patients seen in NHS clinics. They have the potential to reduce time to diagnosis and reduce the cost to the healthcare provider.

To investigate the clinical and cost effectiveness of using home semen analysis tests a randomised controlled trial (RCT) is needed comparing them to laboratory semen analysis (standard care). Before a fully-fledged national trial is planned in a UK setting, the investigators would like to undertake a feasibility study to answer, "Is it feasible to conduct a trial comparing home semen analysis tests with current standard practice for the initial assessment of men referred to the fertility clinic?"

DETAILED DESCRIPTION:
Infertility, defined as the inability to conceive after 12 months of regular unprotected intercourse, is estimated to affect 1 in 7 heterosexual couples, which is an estimated 80 million couples worldwide. Semen analysis, carried out as per the WHO standards in an Andrology laboratory, is the first investigation done for the male partner and reports on multiple semen parameters. Sperm concentration, motility and morphology are the primary reported parameters. Concentration and motility are reported by the laboratory within hours of assessment following sample production, whereas morphology requires extra resources and takes several weeks to produce a report.

Currently, semen analysis requires the patient to attend a hospital clinic, which could be at a significant distance from their home, to produce a sample at a given appointment time that is then analysed by the andrology laboratory without delay. In 30% of UK couples there is an abnormality with at least one semen parameter. The discriminatory ability of semen analysis to distinguish between fertile and infertile men has been questioned, including by the WHO who write the laboratory standards that should be adhered to for examination and processing of human semen.

A systematic review (currently unpublished) of the accuracy of semen analysis as a test of fertility, when undertaken in an Andrology laboratory, concluded that only certain semen parameters in isolation are predictive of reproductive outcomes in treatment-dependent (couples undergoing fertility treatment) and treatment-independent (couples conceiving spontaneously) scenarios. The only parameters predictive of treatment-independent outcomes were sperm concentration and progressive motility. The predictive value of the other semen parameters varied widely between the included studies for treatment-dependent outcomes. Morphology, the most subjectively reported parameter, was only predictive in a population undergoing intrauterine insemination (IUI). However, these studies did not adjust for confounding factors in their statistical analysis and the quality of evidence was low overall.

Despite these findings, semen analysis is an essential component of any fertility work-up and is useful in identifying azoospermia (no sperm present in the sample) and oligozoospermia (low sperm number in the sample). However, a more efficient initial test of male fertility warrants consideration given the limited efficacy of morphology. Home semen analysis tests offer the potential to provide an alternative method for assessment of the male partner and would remove the wide variation in quality control that has been observed between andrology laboratories globally.

Home semen analysis tests can be viewed as a screening tool that provide a simplified, initial assessment of male fertility compared to semen analysis done in an Andrology laboratory, which would be the follow-up diagnostic test if the home test result was abnormal. It could be assumed that the convenience of producing a sample at home in a familiar environment is preferable and no hospital appointment is required. Indeed, a study assessing satisfaction levels of men undergoing laboratory semen analysis who either produced a semen sample at home or in a hospital clinic found significantly higher satisfaction levels by five-point questionnaire in men who produced a sample at home. In addition, a review of men who had undergone a vasectomy reported that 92% would have been more likely to complete post-procedure semen analysis if this could be carried out at home, rather than attending a clinic. This review assessed factors for non-compliance in repeat semen analysis following vasectomy. The primary barriers were noted to be distance, lack of time, and forgetfulness. Home semen analysis tests have the potential to overcome each of these barriers.

Home semen analysis tests are widely available and can be purchased from a local pharmacy or from the internet, but are not currently issued to patients seen in NHS or public sector fertility clinics. Searching a major retailer online and an online search engine resulted in identification of 18 home semen analysis tests that are currently available for purchase, of which 14 are available in the UK. Reported accuracy of the tests available in the UK ranges from 93% to 99%. They all report sperm concentration and six also assess motility. There is no home test available that can analyse morphology.

There are a variety of methods through which home semen analysis tests function. These include an antibody reaction to acrosomal protein SP-10 (a protein specific to male sperm) to produce a test line when a certain threshold of sperm concentration is reached, a colorimetric dye producing a grading of colours depending on the concentration of sperm present, centrifugation to determine the concentration of sperm, and tests that require a smartphone camera to determine both concentration and motility using either a ball lens microscope attachment or a microfluidic chip.

The National Screening Committee specify that a suitable screening test must be "simple, safe, precise, validated and acceptable to the population." They state that the test must have a suitable cut-off level defined and a clear follow-up diagnostic investigation with a positive test result. In addition, one of Wilson and Jungner's (1968) ten principles required in screening for "early disease detection" is that the test should be cost-effective. It is already clear that the follow-up investigation to a home test would be laboratory semen analysis and the cut-off levels used should adhere to those detailed in the WHO laboratory manual. The remaining fundamentals can be viewed in turn when considering the use of a home semen analysis test.

Ten of the home semen analysis tests available for purchase in the UK are CE marked having met the requirements, including for safety, of the section of European Law that governs medical devices. These can therefore be deemed safe to use.

Regarding cost, the mean cost of a single laboratory semen analysis to the NHS was calculated to be £32 in a single centre study based on 2010/2011 data. A more recent publication estimated this cost to be between £46 and £80 in 2018. This varied depending on the Scottish fertility clinic semen analysis was undertaken at and included staff and equipment costs. For a patient paying for semen analysis themselves this ranges from £137.50 in an NHS clinic that also sees self-funded patients (Aberdeen Fertility Centre 2022) to £195 in a private fertility clinic (CARE Fertility 2022).

In comparison, the cost of a home semen analysis test available to purchase in the UK varies from £3.38 per test for a sperm concentration rapid test cassette with 96.6% accuracy to £86.77 (for two tests) for a smartphone-based test reporting motile sperm concentration via a microfluidic chip with 97.8% accuracy. A recent US publication concluded that home semen analysis tests are a "low-cost intervention," which is in agreement with these estimates, and has the benefit of "significantly reduced time to evaluation and treatment for male factor infertility."

Home semen analysis tests have been reported to be accessible for use by patients as minimal or no training is required. Only a single test, the Men's Loupe, which uses a ball lens microscope with a smartphone, requires the user to manually calculate concentration and motility of sperm. The test described is not currently available in the UK. The remaining tests require interpretation of a colour compared to a reference well, the presence or level of a test line, or simply use a smartphone for reporting a result. A study surveying men's opinions after using a home test reported that 92% of men found the test "very easy or easy" to use. There is no published data on the current uptake of home semen analysis tests in the UK by either patients or fertility clinics and this data will be gathered in the feasibility study proposed.

The proposed randomised trial Home semen analysis tests have the potential to reduce the time to diagnosis and reduce the cost to the healthcare provider. To investigate the clinical and cost effectiveness of using home semen analysis tests a randomised controlled trial (RCT) is needed.

To our knowledge, there is no such trial published, but there is one registered (NCT05503862) from the USA - this is an RCT aiming to recruit 200 men with a current female partner attempting to conceive for not more than three months who have not previously had semen analysis. Participants will be randomised to either standard laboratory semen analysis or home semen testing (with the YoSperm® device). Primary outcomes include assessing whether home semen testing was completed, any change in fertility-related WHO-5 wellbeing index, subsequent pursuit of formal male infertility evaluation via a follow-up fertility questionnaire, and any change in fertility-related quality of life.

Before a fully-fledged national trial is planned in a UK setting, the investigators would like to undertake a feasibility study (this protocol). The research plan is described in detail further below. The future trial would randomise men (1:1) to either undergo laboratory semen analysis (standard care) or a home semen analysis test. The reproductive outcomes would be followed up for both arms and compared. The trial is planned to be carried out in a single centre (Aberdeen Fertility Centre).

The following criteria detail the proposed randomised trial at this initial stage and will be further informed by this feasibility study:

* Population: Men with a current female partner aiming to conceive and presenting with infertility
* Intervention: Home semen analysis test (see appendix)
* Comparator: Manual laboratory semen analysis
* Outcome: Live birth
* Time: 12 months

Research plan To assess the feasibility of a randomised trial three work packages (WP) are required. The inclusion criteria for the patient population will be as stated above.

* WP1: Survey of UK clinicians' and scientists' views on home semen analysis tests, including whether a randomised trial is needed to compare them to standard care, and their willingness to recruit to such a trial.
* WP2: Survey of patients' views prior to undergoing routine laboratory semen analysis, including awareness of home testing. Sample size: 100 men.
* WP3: Home testing and post-test survey: Assessment of patients' ability to complete home semen testing with the ExSeed® test, opinions on ease of test use, and views after undergoing both laboratory semen analysis and home testing. Results from the ExSeed® test will be compared to the participant's laboratory semen analysis result to assess the accuracy of the home test. Sample size: 25 men who have undergone WP2 and agreed to trial home testing.

The aim of these work packages is to answer the above research aims and to inform the inclusion and exclusion criteria for the proposed trial. Surveys will be completed electronically, where possible.

ELIGIBILITY:
Work package 1:

Inclusion criterion:

UK fertility specialist, UK embryologist, UK andrology healthcare scientist, or NHS Grampian GP

Exclusion criterion:

Clinical practice is primarily out with the UK

Work package 2:

Inclusion Criteria:

* Male
* Aiming to conceive with a current female partner
* Presenting with infertility
* Laboratory semen analysis at Aberdeen Fertility Centre (standard care) not yet undertaken

Exclusion criteria:

* Younger than 18 years old
* Unable to complete the questionnaire in English
* Current participant in another research study
* Laboratory semen analysis at Aberdeen Fertility Centre already complete

Work package 3:

Inclusion Criteria:

* Male
* Minimum age 18 years old
* Aiming to conceive with a current female partner
* Referred to the fertility clinic with subfertility
* Completed laboratory semen analysis appointment at Aberdeen Fertility Centre
* Smartphone with an operating system of at least Android version 9.0 or iOS version 12.0

Exclusion Criteria:

* Unable to complete the questionnaire in English
* Current participant in another research study
* No valid email address
* Smartphone camera pixel size above 1.4 µm/pixel or below 12 Megapixels
* Attending the clinic for fertility preservation (sperm storage), including men transitioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
What proportion of clinicians are willing to recruit participants to the proposed trial? | 2 months
  Fertility professionals will be asked this in work package 1, which is an online questionnaire. The proposed trial is a randomised controlled trial (RCT) to assess the clinical efficacy of a home semen analysis test versus laboratory semen analysis (standard care).

SECONDARY OUTCOMES:
What is the opinion from clinicians and scientists on the need of such a trial in UK? | 2 months
  Fertility professionals will be asked this in work package 1, which is an online questionnaire.
What is the optimum population, i.e. eligible population for a definitive trial? | 2 months
  Fertility professionals will be asked this in work package 1, which is an online questionnaire.
What are response rates to surveys likely to be in the proposed trial? | 2 months
  This will be assessed in work package 2, which is an online questionnaire.
What proportion of eligible potential participants are willing to be randomised for the proposed trial? | 6 months
  This will be assessed in work package 2 via questionnaire.
What proportion of eligible potential participants are willing to be randomised for the proposed trial following using the home semen analysis test? | 6 months
  This will be assessed in work package 3 with a post-test questionnaire.
What is the optimum primary outcome measure, according to clinicians and scientists, for the proposed trial? | 2 months
  Fertility professionals will be asked this in work package 1, which is an online questionnaire.
Are there any relevant secondary outcome measures that data should also be gathered on for the proposed trial? | 2 months
  Fertility professionals will be asked this in work package 1, which is an online questionnaire.
What duration of follow-up is required to collect outcome data in the proposed trial? | 2 months
  Fertility professionals will be asked this in work package 1, which is an online questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ashleigh C Holt-Kentwell, MBChB, Principal Investigator — University of Aberdeen
Locations (1):
- Aberdeen Fertility Centre, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barratt CL, Mansell S, Beaton C, Tardif S, Oxenham SK. Diagnostic tools in male infertility-the question of sperm dysfunction. Asian J Androl. 2011 Jan;13(1):53-8. doi: 10.1038/aja.2010.63. Epub 2010 Nov 22. PMID 21102478
- [Background] Zegers-Hochschild F, Nygren KG, Adamson GD, de Mouzon J, Lancaster P, Mansour R, Sullivan E; International Committee Monitoring Assisted Reproductive Technologies. The ICMART glossary on ART terminology. Hum Reprod. 2006 Aug;21(8):1968-70. doi: 10.1093/humrep/del171. Epub 2006 Jul 24. PMID 16864610
- [Background] Bjorndahl L, Barratt CLR, Mortimer D, Agarwal A, Aitken RJ, Alvarez JG, Aneck-Hahn N, Arver S, Baldi E, Bassas L, Boitrelle F, Bornman R, Carrell DT, Castilla JA, Cerezo Parra G, Check JH, Cuasnicu PS, Darney SP, de Jager C, De Jonge CJ, Drevet JR, Drobnis EZ, Du Plessis SS, Eisenberg ML, Esteves SC, Evgeni EA, Ferlin A, Garrido N, Giwercman A, Goovaerts IGF, Haugen TB, Henkel R, Henningsohn L, Hofmann MC, Hotaling JM, Jedrzejczak P, Jouannet P, Jorgensen N, Kirkman Brown JC, Krausz C, Kurpisz M, Kvist U, Lamb DJ, Levine H, Loveland KL, McLachlan RI, Mahran A, Maree L, Martins da Silva S, Mbizvo MT, Meinhardt A, Menkveld R, Mortimer ST, Moskovtsev S, Muller CH, Munuce MJ, Muratori M, Niederberger C, O'Flaherty C, Oliva R, Ombelet W, Pacey AA, Palladino MA, Ramasamy R, Ramos L, Rives N, Roldan ER, Rothmann S, Sakkas D, Salonia A, Sanchez-Pozo MC, Sapiro R, Schlatt S, Schlegel PN, Schuppe HC, Shah R, Skakkebaek NE, Teerds K, Toskin I, Tournaye H, Turek PJ, van der Horst G, Vazquez-Levin M, Wang C, Wetzels A, Zeginiadou T, Zini A. Standards in semen examination: publishing reproducible and reliable data based on high-quality methodology. Hum Reprod. 2022 Oct 31;37(11):2497-2502. doi: 10.1093/humrep/deac189. PMID 36112046
- [Background] Bradshaw A, Ballon-Landa E, Owusu R, Hsieh TC. Poor Compliance With Postvasectomy Semen Testing: Analysis of Factors and Barriers. Urology. 2020 Feb;136:146-151. doi: 10.1016/j.urology.2019.10.026. Epub 2019 Nov 26. PMID 31778681
- [Background] Pandey S, McLernon DJ, Scotland G, Mollison J, Wordsworth S, Bhattacharya S. Cost of fertility treatment and live birth outcome in women of different ages and BMI. Hum Reprod. 2014 Oct 10;29(10):2199-211. doi: 10.1093/humrep/deu184. Epub 2014 Jul 24. PMID 25061026
- [Background] Lai JD, Fantus RJ, Meza JA, Hudnall MT, Pham M, Brannigan RE, Ghomrawi HMK, Halpern JA. Cost-effectiveness of Early Screening Home Semen Analysis in Couples Attempting to Conceive. Urology. 2022 Dec;170:104-110. doi: 10.1016/j.urology.2022.06.053. Epub 2022 Sep 14. PMID 36115433
- [Background] Onofre J, Geenen L, Cox A, Van Der Auwera I, Willendrup F, Andersen E, Campo R, Dhont N, Ombelet W. Simplified sperm testing devices: a possible tool to overcome lack of accessibility and inconsistency in male factor infertility diagnosis. An opportunity for low- and middle- income countries. Facts Views Vis Obgyn. 2021 Mar 31;13(1):79-93. doi: 10.52054/FVVO.13.1.011. PMID 33889864
- [Background] Kobori Y. Home testing for male factor infertility: a review of current options. Fertil Steril. 2019 May;111(5):864-870. doi: 10.1016/j.fertnstert.2019.01.032. Epub 2019 Mar 25. PMID 30922654
- [Background] Sommer GJ, Wang TR, Epperson JG, Hatch EE, Wesselink AK, Rothman KJ, Fredriksen LL, Schaff UY, Behr B, Eisenberg ML, Wise LA. At-home sperm testing for epidemiologic studies: Evaluation of the Trak male fertility testing system in an internet-based preconception cohort. Paediatr Perinat Epidemiol. 2020 Sep;34(5):504-512. doi: 10.1111/ppe.12612. Epub 2019 Dec 15. PMID 31838751
- [Background] Gao J, Duan YG, Yi X, Yeung WSB, Ng EHY. A randomised trial comparing conventional semen parameters, sperm DNA fragmentation levels and satisfaction levels between semen collection at home and at the clinic. Andrologia. 2020 Aug;52(7):e13628. doi: 10.1111/and.13628. Epub 2020 May 26. PMID 32458506
- See also: Criteria for appraisal of screening — https://www.bmj.com/content/suppl/2001/04/19/322.7292.986.DC1
- See also: Home Semen Testing in Men Beginning Attempts to Conceive - recruiting study — https://clinicaltrials.gov/ct2/show/study/NCT05503862
- See also: Fertility problems: assessment and treatment NICE Clinical guideline [CG156] — https://www.nice.org.uk/guidance/cg156
- See also: UK government guidance on CE marking — https://www.gov.uk/guidance/ce-marking
- See also: WHO laboratory manual for the examination and processing of human semen Sixth edition — https://www.who.int/publications/i/item/9789240030787